CLINICAL TRIAL: NCT07255300
Title: Follow up Study of the Effects of the Longevity and the Fasting Mimicking Diet on Body Composition, Age-related Risk Factors and Biomarkers of Aging in a Randomized Study 1 and 2
Brief Title: Follow up Study of Varapodio Trial: Effect of Longevity and Fasting Mimicking Diet on Risk Factors Age Correlated and Biomarkers of Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Valter Longo (Other)
Collaborators: Universita degli Studi di Palermo (Other); University of Calabria (Other); Regione Calabria / Comune Varapodio (Unknown); European Longevity Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2025-08-21; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-08

CONDITIONS: Fat Mass; Risk Factors Cardiovascular Disease; Epigenetic Aging; Metabolism Changes; Overweight (BMI > 25); Risk Behavior; Obesity (Disorder)
Keywords: fasting; fasting mimicking diet; Longevity Diet; Longevity; Diet; Aging; FMD; Nutrition; Diseases; LD; Clinical Trial; Randomized; Health; Fat Mass
MeSH Terms: conditions — Overweight; Risk-Taking; Obesity; Fasting; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting Mimicking Diet (Experimental): The fasting-mimicking diet (FMD) group, will be instructed on the benefits and use of the fasting-mimicking diet and how it should be used. This group will have to perform the fasting-mimicking diet once every 4 months (3 cycles in 1 year).
  Interventions: Behavioral: fasting mimicking diet

INTERVENTIONS:
Behavioral: fasting mimicking diet — The subjects will be instructed to follow their usual diet plan, except for 5 days when they eat the foods in the FMD box.The fasting-mimicking diet consists of a blend of 100% plant based nutrients generally regarded as safe. The formulation of these products is based on studies carried out at the Longevity Institute of the University of Southern California and his collaborators over several decades of studies.
  This food plan provides for the replacement of the normal diet with the organic plant products contained in the fasting-mimicking diet for five consecutive days.

SUMMARY:
A large ongoing randomized, open-label trial aimed at evaluating the effects of two different dietary interventions, FMD and LD, on body composition and cardiovascular (CV) biomarkers in a real word population (NCT05698654) is actually ongoing. This trial started in January 2024 will enrol 501 adult subjects between the ages of 30 and 65: 167 subjects randomized to the FMD arm with a 5-day meal program once every three months for a 6-month period (arm 1); 167 subjects randomized to follow the FMD plus a Longevity Diet program (FMD+LD) for a 6-month period (arm 2); 167 randomized to the control group (arm 3) that will continue their usual diet. On 2024,410, participants were enrolled and randomly assigned to FMD, FMD + LD, or control arm. Although preliminary data demonstrated the beneficial effects of such nutritional plans on body weight, BMI, body composition, and cardiovascular (CV) biomarkers, limited data is available on the long-term effects of these powerful nutritional interventions.

DETAILED DESCRIPTION:
Background Information With a growing aging population all over the world, healthy ageing is an important goal for public health.

Dietary restriction (DR), implemented as chronic and coordinate reduced intake of all dietary constituents except vitamins and minerals, was first shown more than 80 years ago to extend lifespan in model organisms and in humans. Dietary interventions that avoid unrealistic levels of self-deprivation, and pharmacological interventions that recapture beneficial effects of DR, are therefore important goals to improve human health during aging. Despite its potential for disease prevention and treatment, prolonged fasting is difficult to implement in human subjects and may exacerbate preexisting nutritional deficiencies, making it not feasible and/or safe for children, the elderly, frail individuals, and even most of the healthy adults. Fifteen years of extensive preclinical and clinical studies sponsored by the National Institutes of Health (NIH) and conducted at the Longevity Institute and Diabetes and Obesity Research Institute of the University of Southern California (USC) resulted in the development of a very promising dietary interventions effective in extending not only longevity but also the healthy life span: the fasting mimicking dietâ (FMD).

Fasting Mimicking Diet The fasting-mimicking diet (FMD) is a 5-day meal program to be consumed every 1 to 6 months based on an authorized healthcare professional's recommendation. It is designed to promote the body's natural ability to protect, regenerate and rejuvenate itself. In clinical studies, FMD has been shown to reduce abdominal fat and maintain healthy levels of blood glucose, C-reactive protein (CRP), and insulin-like growth factor 1 (IGF-1) (Wei et al., 2017). Well-designed clinical trials, such as the study conducted by Houston et al. utilizing an independent review board (IRB) approved protocol, have demonstrated the safety and short-term benefits of plant-based nutraceuticals and food restriction in individuals with chronic hypertension (Houston et al., 2014).

A large ongoing randomized, open-label trial aimed at evaluating the effects of two different dietary interventions, FMD and LD, on body composition and cardiovascular (CV) biomarkers in a real word population (NCT05698654) is actually ongoing. This trial started in January 2024 will enrol 501 adult subjects between the ages of 30 and 65: 167 subjects randomized to the FMD arm with a 5-day meal program once every three months for a 6-month period (arm 1); 167 subjects randomized to follow the FMD plus a Longevity Diet program (FMD+LD) for a 6-month period (arm 2); 167 randomized to the control group (arm 3) that will continue their usual diet. On 2024,410, participants were enrolled and randomly assigned to FMD, FMD + LD, or control arm. Although preliminary data demonstrated the beneficial effects of such nutritional plans on body weight, BMI, body composition, and cardiovascular (CV) biomarkers, limited data is available on the long-term effects of these powerful nutritional interventions.

The objective of the study is to determine long-term trends of a 5-day FMD meal program in patients already subjected to FMD in a previous trial (NCT05698654) and that will continue an FMD-based plan to assess its long-term effect on fat mass maintenance. The secondary objectives are to determine long-term trends of a 5-day FMD meal program in patients already subjected to FMD who will continue an FMD-based plan to assess its long-term effect on the maintenance of body weight, body mass index, blood pressure, IGF-1, haemoglobin A1c, fasting glucose, LDL, total cholesterol, C-Reactive Protein, and the proportion of participants who received medications at baseline.

Primary endpoint: maintenance of at least 50% of the fat mass lost during the previous trial and measured after one follow up year on FMD every 3 months Secondary endpoints: maintenance of at least 50% of one or more risk factors improvements achieved during the previous clinical trial and measured after one year of follow up FMD cycles every 3 months including improvements in: body mass, body mass index, blood pressure, IGF-1, haemoglobin A1c, fasting glucose, LDL, total cholesterol, and C-Reactive Protein. Determine long-term trends in the reduction/stabilization in the use of antihypertensive and glucose-lowering drugs or other commonly used medications.

Follow up clinical trial including participants of the approved studies "Studio degli effetti della dieta mima-digiuno e della dieta della longevità sulla composizione corporea, fattori di rischio per malattie età-correlate e marcatori dell'invecchiamento in uno studio randomizzato" and "Studio degli effetti della dieta mima-digiuno e della dieta della longevità sulla composizione corporea, fattori di rischio per malattie età-correlate e marcatori dell'invecchiamento in uno studio randomizzato-2" that will follow 5-day of the FMD meal program every three months, for one year.

Selection and withdrawal of subjects of the previous clinical study

The participants will be identified within the intervention groups of the previous clinical studies (Studio degli effetti della dieta mima-digiuno e della dieta della longevità sulla composizione corporea, fattori di rischio per malattie età-correlate e marcatori dell'invecchiamento in uno studio randomizzato1 and 2) who are willing to start a new study for other 12 months, and who completed the study less than 6 months prior to starting the new study and achieved the study's objectives. Blood tests and a nutritional assessment will be conducted, serving as the baseline for the new study. The recruitment period will last up to 3 years

The assessment schedule lists all the assessments and when they are to be performed.

Potential participants already subjected to a 5-day fasting-mimicking diet (FMD) program either alone or in combination with the longevity diet previously enrolled in one of the two interventional arms and who completed the clinical study NCT05698654 less than three months before the enrolment period will be contacted via telephone to determine preliminary eligibility and interest. Once participants meet all inclusion/exclusion criteria, they will be offered by study staff the opportunity to learn more about the research opportunity before any procedure is performed. Participants meeting eligibility will be then invited to attend a baseline and two follow-up visits

Participants will be given three boxes of FMD together with ketone test strips to self-monitor urinary ketone bodies during the FMD cycles. Detailed information on the FMD plans will be also given during the visit. Baseline visit will also include body composition assessment using Bioelectrical Impedance Analysis (BIA), measurement of height, weight, and vital signs, medical history, current medications and a collection of fasting blood for the genetic analysis (25 mL: 7.5 mL for serum, 7.5 mL for plasma, 10 mL for white blood cells).

The follow-up visits will be carried out after three (follow-up visit 1) and five (follow-up visit 2) FMD cycles (6 and 12 months), in order to evaluate the progress of the trial.

Follow-up visit 1 During the first follow-up visit, the study staff will assess the signs and symptoms of adverse events and review compliance to the FMD program. The visit will also include body composition assessment using BIA, measurement of height, weight, and vital signs, medical history and current medications. Participants will receive the FMD boxes for the remaining two cycles together with the ketone test strips for self-monitoring of urinary ketone bodies during the FMD cycles.

During the second follow-up visit, the study staff will assess the signs and symptoms of adverse events and review compliance to the FMD program. This visit will also include body composition assessment using BIA, measurement of height, weight, and vital signs, medical history and current medications. In addition, a collection of fasting blood for haematological and for the genetic analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

Subjects of 30-65 years of age;

Exclusion Criteria:

individuals with a family member already included in the study; individuals who are allergic to tree nuts (macadamia, cashew, almond, pecan), soy, oats, sesame, or celery/celeriac; pregnant females; Individuals with any documented cancer diagnosis within the past 5 years; documented myocardial infarction within past 5 years; documented cerebrovascular accident within past 5 years; chronic steroid use (longer than 45 consecutive days); insulin-dependent diabetes mellitus; individuals taking insulin or insulin-like drugs and individuals taking hypoglycemic agents other than metformin. In this last case, close attention will therefore be paid to the self-monitoring of blood glucose during the FMD cycles; Individuals with severe hypertension (systolic greater than 200 mmHg and or diastolic greater than 105 mmHg.

Change in prescription medications, over-the-counter (OTC) medications, medical foods, and nutritional supplements within 30 days prior to the start and for the duration of the study.

Use of medications classified as narcotics 15 days prior start and for the duration of the study.

Use of prescription medications and/or over-the-counter medications for acute and semi- acute medical conditions 15 days prior to start and for the duration of the study.

Use of acetaminophen is permitted on an as-needed basis. Use of an investigational drug or participation in an investigational study within 30 days prior to the start and for the duration of the study.

Use of oral or injectable corticosteroids within 30 days prior to the start and for the duration of the study.

Use of anticoagulant medications (heparin compounds or warfarin) within 30 days prior to the start and for the duration of the study. Use of aspirin 81 mg or 325 mg once daily is permitted.

Use of neuroactive prescription medications including major and atypical antipsychotic medications, anti-depressants, anti-anxiolytics, and epilepsy medications within 30 days prior to the start and for the duration of the study.

(subjects will not be allowed to discontinue prohibited prescription medications to meet enrolment criteria).

A history of allergy or intolerance to study products. Detailed descriptions of study product are included in Section 4.1 and 4.2, appended to the Study Informed Consent.

Clinically significant vital sign abnormalities (systolic blood pressure <90 mmHg or >200 mmHg, diastolic blood pressure <50 mmHg or >105 mmHg or resting heart rate of <50 or >100 bpm) at screening visit.

A serious, unstable illness including cardiac, hepatic, renal, gastrointestinal, respiratory, endocrinologic, neurologic, immunologic, or hematologic disease.

Known infection with HIV, TB or Hepatitis B or C.

A current diagnosis or personal history of:

Any cardiovascular disease including myocardial infarction, angina, cardiovascular surgery (within 5 years), congestive heart failure, cardiac arrhythmias or conduction abnormalities, cerebrovascular accident, transient ischemic attack (TIA), or peripheral vascular disease, deep vein thrombosis or pulmonary embolus. Diabetes mellitus requiring inhaled or injected insulin.

Any autoimmune disease such as inflammatory bowel disease (including Crohn's disease and/or ulcerative colitis), multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus, polymyositis, scleroderma and/or thyroiditis.

Any significant liver or kidney disease such as cirrhosis or non-alcoholic fatty liver disease, glomerulonephritis, and/or ongoing dialysis treatment.

Any malignancy (with the exception of adequately treated malignancies with no known recurrence for >2 years).

Any serious mental illness including a history of attempted suicide. Any medical condition that in the opinion of the primary care doctor or a specialist would preclude safe participation in this study or interfere with compliance.

Use of drugs of abuse (such as marijuana, cocaine, phencyclidine [PCP] and methamphetamine) 15 days prior to Day 1 and for the duration of the study.

History of regular intake of >14 alcoholic drinks per week for females, and >21 drinks per week for males (1 drink = 35 cl. beer, 12 cl. wine, or 30 ml. hard liquor).

Technical reasons

Any condition in which bioelectrical impedance testing would be impossible or uninterpretable (e.g. prostheses in extremities on both sides, limb amputation, implanted pacemaker, inability to lay still or supine, or skin defects on preferred electrode placement sites.

Other Exclusion Criteria: Inability to comply with study and/or follow-up visits.

Any concurrent condition (including clinically significant abnormalities in medical history, physical examination or laboratory evaluations) which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.

Any sound medical, psychiatric and/or social reason which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.

Abnormal laboratory findings including: abnormal blood counts (hematocrit < 33% or > 47%; WBC < 3.0 or > 12.0 x10^3/mm3; platelets < 140 or > 500 x 10^9/L); abnormal kidney function test (creatinine > 2.5 mg/dL) or liver function test(s) (AST, ALT, alkaline phosphatase) > 1.5X the upper limit of normal; serum calcium > 11 mg/dL); serum K < 3.5 mEq/L; Na < 134 or > 148 mmolL-1 Women of Childbearing Potential Contraception: the effects of the study products on the developing human fetus have not been studied extensively. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Females of childbearing potential will have a pregnancy test prior to receiving study products. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform study staff and her primary care physician immediately.

Pregnancy: because there is an unknown but potential risk for adverse events in pregnant women during treatment with the study products, pregnant women are not eligible for study participation.

Breast-feeding: Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study products, breastfeeding mothers are not eligible for study participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-05-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Body Fat Percentage | Time Frame: Comparison of the clinical marker up to 7 days after the randomization and 1 year after the randomization.
  Maintenance of at least 50% of the fat mass lost during the previous trial and measured after one follow up year on FMD every 3 months.

SECONDARY OUTCOMES:
maintenance of at least 50% of one or more risk factors improvements achieved during the previous clinical trial | comparison from day 1 after randomization and one year after the randomization
  maintenance of at least 50% of one or more risk factors improvements achieved during the previous clinical trial and measured after one year of follow up FMD cycles every 3 months including improvements in: body mass, body mass index, blood pressure, IGF-1, haemoglobin A1c, fasting glucose, LDL, total cholesterol, and C-Reactive Protein. Determine long-term trends in the reduction/stabilization in the use of antihypertensive and glucose-lowering drugs or other commonly used medications.

CONTACTS AND LOCATIONS:
Overall Officials: Romina Inés Cervigni, Study Director — Fondazione Valter Longo; Alberto Montesanto, Study Chair — University of Calabria
Locations (1):
- Ambulatorio Medico presso Biblioteca Comunale, Varapodio, Calabria, Italy, Italy

REFERENCES:
- [Result] Pollack MN. Insulin, insulin-like growth factors, insulin resistance, and neoplasia. Am J Clin Nutr. 2007 Sep;86(3):s820-2. doi: 10.1093/ajcn/86.3.820S. PMID 18265475
- [Result] Levine ME, Suarez JA, Brandhorst S, Balasubramanian P, Cheng CW, Madia F, Fontana L, Mirisola MG, Guevara-Aguirre J, Wan J, Passarino G, Kennedy BK, Wei M, Cohen P, Crimmins EM, Longo VD. Low protein intake is associated with a major reduction in IGF-1, cancer, and overall mortality in the 65 and younger but not older population. Cell Metab. 2014 Mar 4;19(3):407-17. doi: 10.1016/j.cmet.2014.02.006. PMID 24606898
- [Result] Wei M, Brandhorst S, Shelehchi M, Mirzaei H, Cheng CW, Budniak J, Groshen S, Mack WJ, Guen E, Di Biase S, Cohen P, Morgan TE, Dorff T, Hong K, Michalsen A, Laviano A, Longo VD. Fasting-mimicking diet and markers/risk factors for aging, diabetes, cancer, and cardiovascular disease. Sci Transl Med. 2017 Feb 15;9(377):eaai8700. doi: 10.1126/scitranslmed.aai8700. PMID 28202779
- [Result] Gallus S, Odone A, Lugo A, Bosetti C, Colombo P, Zuccaro P, La Vecchia C. Overweight and obesity prevalence and determinants in Italy: an update to 2010. Eur J Nutr. 2013 Mar;52(2):677-85. doi: 10.1007/s00394-012-0372-y. Epub 2012 May 27. PMID 22645105
- [Result] Houston M, Hays L. Acute effects of an oral nitric oxide supplement on blood pressure, endothelial function, and vascular compliance in hypertensive patients. J Clin Hypertens (Greenwich). 2014 Jul;16(7):524-9. doi: 10.1111/jch.12352. Epub 2014 Jun 24. PMID 24962851
- [Result] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889
- [Result] Knoops KT, de Groot LC, Kromhout D, Perrin AE, Moreiras-Varela O, Menotti A, van Staveren WA. Mediterranean diet, lifestyle factors, and 10-year mortality in elderly European men and women: the HALE project. JAMA. 2004 Sep 22;292(12):1433-9. doi: 10.1001/jama.292.12.1433. PMID 15383513

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT07255300/Prot_ICF_000.pdf